CLINICAL TRIAL: NCT03961022
Title: Effects of Dietary Supplementation With ReWin(d) on the Recovery of Young Athletes Suffering From Delayed-Onset Muscle Soreness Induced by Acute Exercice: A Pilot Randomized, Double-blind, Placebo Controlled Trial
Brief Title: Effects of ReWin(d) Supplementation on the Recovery of DOMS Induced by Acute Exercice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Natural Origins (Industry)
Collaborators: European University of Madrid (Other)
Responsible Party: Principal Investigator, Margarita Pérez Ruiz, Principal Investigator. Full Profesor in Physical Activity and Sport. Exercise physiology., European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Nat.Origins-ReWin(d)-2019
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Muscle Soreness; Delayed-onset Muscle Soreness
Keywords: DOMS; Fatigue rate; Heart rate variability; Pain; Jump performance
MeSH Terms: conditions — Myalgia; Pain

STUDY DESIGN:
Intervention Model Description: Single dose, Randomized, Double Blinded, Placebo-controlled Study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReWin(d) (Active Comparator): Subjects have to take ReWin(d) capsules (3 times a day, total 2 g/day) during breakfast, lunch and diner, during 4 weeks + 3 days after acute exercice
  Interventions: Dietary Supplement: Polyherbal supplement: ReWin(d) vs Placebo
- placebo (Placebo Comparator): Subjects have to take Placebo capsules (3 times a day, total 2 g/day) during breakfast, lunch and diner, during 4 weeks + 3 days after acute exercice
  Interventions: Dietary Supplement: Polyherbal supplement: ReWin(d) vs Placebo

INTERVENTIONS:
Dietary Supplement: Polyherbal supplement: ReWin(d) vs Placebo — Supplementation during 4 weeks + 72 hours post acute exercice

SUMMARY:
The study will assess the recovery and performance of young athletes suffering from muscle damage induced by physical exercise. Model by comparing the safety and efficacy of ReWin(d) supplemention during 4 weeks to placebo over 72 hours post exercice.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo controlled, parallel group, pilot safety and efficacy study.

40 healthy young male athetes were randomly assigned to the ReWin(d) or Placebo group. After 4 weeks supplementation (either 2 g daily of ReWin(d) capsules or placebo capsules). the participants were subjected to a 1 hour plyometric exercise session to induce DOMS. At 0 hours, 24 hours, 48 hours and 72 hours post exercise, the volunteers have been assessed to determine: (i) pain perception, (ii) fatigue rate, (iii) sport performance (effectiveness of a jump) and (iv) muscle damage and inflammation by I-R thermography and biomarkers

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Young athletes
* Training at least 3 times per week
* Agree not to initiate any new exercise or diet programs during the entire study period
* Agree not to change their current diet or exercise program during the entire study period
* Agree not to stretch, utilize ice massage, take anti-inflammatory medications (eg, aspirin, ibuprofen), or use any other treatment for the duration of the trial.

Exclusion Criteria:

* Previous history of upper extremity injury or knee joint pain
* Use of anti-inflammatory medications or pain medications 1 week before the screening visit and during the study
* Daily use of dietary supplements and herbal supplements beginning at the screening visit and during the study
* Antibiotic use in past 3 months
* Chronic disease

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Effects of ReWin(d) on muscle recovery induced by physical exercise | Change from baseline at 0 hours, 24 hours, 48 hours and 72 hours post plyometric exercises session to induce DOMS
  Sport performance (effectiveness of a jump) after exercise-induced muscle damage

SECONDARY OUTCOMES:
Effects of ReWin(d) on muscle damage induced by physical exercise | Change from baseline at 0 hours, 24 hours, 48 hours and 72 hours post plyometric exercises session to induce DOMS
  Muscle skin temperature monitored by IR-camera.
Effects of ReWin(d) on pain perception induced by physical exercise | Change from baseline at 0 hours, 24 hours, 48 hours and 72 hours post plyometric exercises session
  Visual Analogue Scale pain perception after exercise-induced muscle damage
Effects of ReWin(d) on fatigue rate induced by physical exercise | Change from baseline at 0 hours, 24 hours, 48 hours and 72 hours post plyometric exercises session
  Heart Rate Variability assessment after exercise-induced muscle damage
Effects of ReWin(d) on Gut Microbiota | Change from baseline dose after 4 weeks of intervention
  Determination of Microbiota composition by 16S rRNA Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez Ruiz, MD(Res), Principal Investigator — European University of Madrid
Locations (1):
- European University of Madrid, Villaviciosa de Odón, Madrid, Spain

REFERENCES:
- [Derived] Dominguez-Balmaseda D, Diez-Vega I, Larrosa M, San Juan AF, Issaly N, Moreno-Perez D, Burgos S, Sillero-Quintana M, Gonzalez C, Bas A, Roller M, Perez-Ruiz M. Effect of a Blend of Zingiber officinale Roscoe and Bixa orellana L. Herbal Supplement on the Recovery of Delayed-Onset Muscle Soreness Induced by Unaccustomed Eccentric Resistance Training: A Randomized, Triple-Blind, Placebo-Controlled Trial. Front Physiol. 2020 Jul 21;11:826. doi: 10.3389/fphys.2020.00826. eCollection 2020. PMID 32848820